CLINICAL TRIAL: NCT01142206
Title: The Effects of Two Different Leisure-time Activity Prescriptions on Eating and Activity Behaviors During Behavioral Weight Loss Treatment
Brief Title: The Leisure-time Activity and Nutrition Program
Acronym: LEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7521B
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Leisure-time activities; Physical Activity; Television watching; Dietary Intake; Energy; Behavioral; Healthy Eating
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity; Behavior | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Active Comparator): A standard behavioral weight loss intervention with a physical activity prescription of 200 minutes of moderate intensity physical activity per week.
  Interventions: Behavioral: Dietary; Behavioral: Physical Activity
- Physical Activity & TV Watching (Experimental): A standard behavioral weight loss intervention with a physical activity prescription of 200 minutes of moderate intensity physical activity per week and an additional prescription of reducing TV watching to 10 hours per week or less.
  Interventions: Behavioral: Dietary; Behavioral: Physical Activity; Behavioral: TV Watching + Physical Activity

INTERVENTIONS:
Behavioral: Dietary — All participants in the investigation will receive a standard 8-week behavioral obesity intervention with 8 weekly, 1 hour group counseling and education sessions. The intervention will include a reduced caloric prescription (1200-1500 kcal/day) and fat gram prescription (30% or less kcals from fat).
Behavioral: Physical Activity — All participants will receive a physical activity goal of 200 minutes/week of moderate-intense physical activity.
Behavioral: TV Watching + Physical Activity — The TV Watching + physical activity arm will receive a TV watching goal of watching less than 10 hours of TV/week.
  Arms: Physical Activity & TV Watching

SUMMARY:
The purpose of this investigation is to conduct an 8-week pilot study to examine the effects of two different leisure-time activity prescriptions on dietary intake, leisure-time activities, and weight loss in 30 adults receiving an 8-week behavioral weight loss intervention.

DETAILED DESCRIPTION:
In adult observational studies, TV viewing has been positively related to overweight and obesity. It is theorized that TV watching influences eating and activity behaviors, such that with greater TV watching less physical activity and greater consumption of energy occurs, producing a positive energy balance state. While no experimental research has been conducted with adults examining the influence of reducing TV watching on weight status, experimental research conducted with children does indicate that lower levels of TV watching can produce reduced energy intake and greater levels of physical activity. Most importantly, family-based, behavioral childhood obesity interventions that have targeted reducing sedentary behaviors (which includes TV watching) have found that as compared to targeting increasing physical activity during treatment, similar increases in activity and fitness occur, but that greater weight loss and greater increases in liking for physical activity occur when sedentary behaviors, as compared to physical activity, are targeted in family-based behavioral childhood weight control programs.

All participants in the investigation will receive a standard 8-week behavioral obesity intervention. The intervention will include a reduced caloric prescription (1200-1500 kcal/day) and fat gram prescription (30% or less kcals from fat). One condition will receive an activity goal (200 minutes/week of moderate-intense physical activity [Physical Activity]), while the other condition will receive a TV watching goal (10 hours/week) and a physical activity goal (200 minutes/week of moderate-intense physical activity [TV + Physical Activity]. Participants will be assessed at 0 and 9 weeks (pre- and post-intervention) on measures of dietary intake, physical activity, TV watching, time-use, motivation, liking of physical activity and TV watching, and weight.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 45 kg/m2
* Watch > 16 hours per week of TV
* Engage in < 100 minutes of moderate-intense physical activity per week

Exclusion Criteria:

* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q).
* Individuals self-reporting joint problems, prescription medication usage related to heart conditions, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
* Report being unable to walk for 2 blocks (1/4 mile) without stopping.
* Report no TVs in the home or 5 or more TVs in the home viewed by the participant (TVs in participant's children's bedrooms will not be counted)
* Are unwilling to have TV Allowances attached to TVs in the home.
* Report other household members are unwilling to use the TV Allowance.
* Report major psychiatric diseases or organic brain syndromes via a phone screen.
* Are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months.
* Are currently participating in a program to increase physical activity and/or decrease TV watching time.
* Intend to move to another city within the time frame of the investigation.
* Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation.
* Have had gastric surgery for weight loss.
* Are unwilling to attend weekly sessions.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Time spent in moderate-intensity physical activity | Week 9
  Participants will be given a closed motion sensor (Omron HJ-720 ITC Pocket Pedometers) to wear over the course of the program to measure number of steps and time spent engaged in moderate -intensity and higher physical activity. Days in which the sensor has been worn at least 10 hours only will be counted towards the seven days. The motion sensors will be downloaded onto computers at the baseline assessments and at week 9. During weeks 0 and 9 all participants will also keep a record of the self-reported physical activity.
Television watching time | Week 9
  TV monitoring devices ("TV Allowances") will be hooked onto participants' home TVs by research staff. The devices will record the number of hours per week of TV the research participant is watching. Participants will also be asked to keep a record of their self-reported TV watching at 0 and 9 weeks.

SECONDARY OUTCOMES:
Liking of physical activity and TV watching | Week 9
  Participants will rate the pleasantness of engaging in physical activity and TV watching using a 100 mm visual analogue scale (VAS), anchored on the left with "very unpleasant" and on the right by "very pleasant."
Motivation for physical activity | Week 9
  Motivation for physical activity willbe measured via severl previously validated questionnaires.
Dietary Intake (calories and % calories from fat) during TV watching or computer use | Week 9
  Dietary intake will be assessed by three-day food records at weeks 0 and 9. Along with recording foods and drink consumed, participants will indicate in the record when TV is being watched as food and drinks are consumed. These food records will be reviewed to ensure that information written about consumption is complete and incomplete dairies will be reviewed with participants. Dietary data will be analyzed using NDS-R software.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, RD, LDN, Principal Investigator — University of Tennessee; David Bassett Jr., PhD, Study Chair — University of Tennessee; Dixie Thompson, PhD, Study Chair — University of Tennessee; Amy Gorin, PhD, Study Chair — University of Connecticut
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States

REFERENCES:
- See also: This is the website for the Healthy Eating and Activity Laboratory (HEAL), where this program is being conducted.) — http://heal.utk.edu/